CLINICAL TRIAL: NCT05565066
Title: A Real-world Comparison of FNB and FNA in IHC-required Lesions: A Prospective, Multicenter Study.
Brief Title: A Real-world Comparison of FNB and FNA in IHC-required Lesions.
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Bin Cheng, Dr., Huazhong University of Science and Technology
Other Study IDs: FNB-2022tj
Record Dates: First submitted 2022-09-26; First posted 2022-10-04 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Neuroendocrine Tumors; Autoimmune Pancreatitis; Gastrointestinal Stromal Tumors
Keywords: Endoscopic ultrasound; Pathological diagnosis; Fine needle aspiration; Fine needle biopsy
MeSH Terms: conditions — Neuroendocrine Tumors; Autoimmune Pancreatitis; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FNB group: FNB needles adpted to acquire lesion tissues according patients' advice and patients' willings.
  Interventions: Device: FNB group
- FNA group: FNA needles adpted to acquire lesion tissues according patients' advice and patients' willings.
  Interventions: Device: FNA group

INTERVENTIONS:
Device: FNB group — Fine-needle-biopsy (Echotip ProCore Needle)
  Groups: FNB group
Device: FNA group — Fine-needle-aspiration (Echotip Needle)
  Groups: FNA group

SUMMARY:
Endoscopic ultrasound (EUS)-guided fine needles with side fenestrations are used to collect aspirates for cytology analysis and biopsy samples for histologic analysis. The investigators conducted a large, multicenter study to compare the accuracy of diagnosis via specimens collected with fine-needle biopsy (FNB) versus fine-needle aspiration (FNA) for patients with lesions requiring immunohistochemistry (IHC) pathological diagnosis.

DETAILED DESCRIPTION:
Current guidelines recommend FNA and FNB needles equally for pancreatic and other deep-seated lesions. However, some studies indicate that the sample adequacy for histologic evaluation is higher when using FNB compared with FNA needles. The diagnosis of neuroendocrine tumor (NET), autoimmune pancreatitis (AIP), and other gastrointestinal stromal tumors require high-quality tissue sampling for IHC diagnosis. Whether FNB is superior to FNA in these IHC-required lesions remains unclear.

The investigators performed this at 2 tertiary care centers in China. The study prospectively collected patients undergoing EUS for a solid mass (>1 cm) in the pancreas, abdomen, mediastinum, or pelvic cavity from December 2014 diagnosed with AIP, NET, mesenchymal tumors, and Lymphoma. Patients accepted FNB or FNA according to doctors' and patients' willingness in a real-world setting. All procedures were performed by experienced endosonographers; cytologists and pathologists were blinded to the sample collection method. Patients were followed for at least 48 weeks, and final diagnoses were obtained after surgery, imaging analysis, or resolution of the lesion. The primary aim was to compare diagnostic yields of EUS-FNA with EUS-FNB for all solid masses, then separately as AIP, NET, mesenchymal tumors, and lymphoma. The secondary endpoint was the quality of the histologic specimen.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years;
* presence of a solid mass lesion was confirmed by at least 1 imaging modality and it was located within pancreas, abdomen, mediastinum, or pelvic cavity;
* mass size >1 cm;
* final diagnoses were obtained after surgery, imaging analysis, or resolution of the lesion, including AIP, NET, mesenchymal tumors, and lymphoma.

Exclusion Criteria:

* coagulopathy (international normalized ratio, 1.5);
* thrombocytopenia (platelet count <50,000/mm3);
* acute pancreatitis within the previous 2 weeks;
* inability to safely perform EUS-TA (eg, cardiorespiratory dysfunction, mental diseases, or drug addiction);
* refusal or inability to provide an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yields of EUS-FNA with EUS-FNB for solid masses | From admission until the date of pathological diagnosis obtained or follow-up up to 24 months
  Overall dignostic yields of all solid lesions
Diagnostic yields of EUS-FNA with EUS-FNB for solid masses | From admission until the date of pathological diagnosis obtained or follow-up up to 24 months
  dignostic yields of AIP
Diagnostic yields of EUS-FNA with EUS-FNB for solid masses | From admission until the date of pathological diagnosis obtained or follow-up up to 24 months
  dignostic yields of NET
Diagnostic yields of EUS-FNA with EUS-FNB for solid masses | From admission until the date of pathological diagnosis obtained or follow-up up to 24 months
  dignostic yields of GIST

SECONDARY OUTCOMES:
Quality of histologic specimen | From admission until specimen evaluted by two independent pathologists, assessed up to 4 weeks
  Specimen adequacy - whether adequate for IHC staining
Quality of histologic specimen | From admission until specimen evaluted by two independent pathologists, assessed up to 4 weeks
  Specimen adequacy - tissue intergrity

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, HUST, Wuhan, Hubei, China